CLINICAL TRIAL: NCT06413810
Title: A Randomised, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Effects of a Food Ingredient on Self-reported Stress in Healthy Adults
Brief Title: The Effects of a Food Ingredient on Self-reported Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-177
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food ingredient (Experimental): Standard food ingredient under investigation
  Interventions: Other: Calmarell
- Placebo (Placebo Comparator): Matched standard food ingredient with no impact
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Calmarell — Food ingredient
  Arms: Food ingredient
Other: Placebo — Blinded placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate if a food ingredient can improve stress in healthy adults who experience moderate symptoms of self-reported stress. The main question it aims to answer is if 4 weeks of daily intake of the ingredient reduces stress compared to 4 weeks of daily intake of a placebo product.

Participants will:

* consume both the test and placebo products for 4-weeks each in a randomised order, with 4 weeks in between
* visit the test site 6 times over the 13 weeks
* complete a series of assessments on stress and sleep quality and provide blood, stool and saliva samples

DETAILED DESCRIPTION:
A double-blind, randomised, placebo-controlled, crossover study with 6 visits over 13-weeks. Participants will consume study product or placebo for two 4-week intervention periods.

Primary Objective: To evaluate in healthy adults, experiencing moderate symptoms of self-reported stress, the effect of 4-week daily supplementation of a food ingredient versus placebo on stress.

Secondary Objectives: To evaluate in healthy adults, experiencing moderate symptoms of self-reported stress, the effect of 4-week daily supplementation of a food ingredient versus placebo on:

* Mood
* Plasma GABA levels
* Salivary cortisol awakening response (CAR)
* Acute effects on stress
* Faecal GABA

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, the Participant must fulfil all the following criteria:

  1. Be able to give written informed consent.
  2. Be between 18 and 50 years of age.
  3. Has a BMI between ≥ 18.0 and ≤ 30.0 kg/m2.
  4. Have moderate stress, as measured on Cohen's Perceived Stress Scale (PSS), with a score between 14 and 26 (inclusive) at both Screening and Baseline Visits.
  5. Is in general good health, as determined by the investigator.
  6. Willing to consume the Study Product daily for the duration of the study and comply with the study procedures.

Exclusion Criteria:

* The presence of any of the following criteria will exclude the Participant from participating in the study:

  1. Scores ≥10 on General Anxiety Disorder 7 item (GAD-7) questionnaire.
  2. Scores ≥10 Patient Health Questionnaire 9 item (PHQ-9).
  3. Participants who are pregnant or wish to become pregnant during the study.
  4. Participants who are lactating and/or currently breastfeeding.
  5. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

     1. Complete abstinence from intercourse two weeks prior to administration of the study product, throughout the human study, until the completion of follow-up procedures or for two weeks following discontinuation of the study product in cases where Participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
     2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that Participant.
     3. Sexual partner(s) is/are exclusively female.
     4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.
     5. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
  6. Is hypersensitive to any of the components of the Study Product.
  7. Have a significant acute or chronic coexisting illness such as such as uncontrolled hypertension, type 1 or 2 diabetes, cardiovascular diseases or any condition which may, in the opinion of the investigator, impact their ability to participate in the study or impact the study outcomes.
  8. Use of systemic antibiotics within the 12 weeks prior to Visit 1.
  9. Use of systemic immunosuppressant drugs, steroids, etc. within the 12 weeks prior to Visit 1.
  10. Participants diagnosed and treated with prescribed medications for anxiety and depression in the 12 weeks prior to Visit 1.
  11. Participants who have taken 3 doses laxative or anti-diarrheal medication in the past 12 weeks, at investigator discretion.
  12. Herbal treatments for mood disorders or psychological conditions (e.g., valerian, St. John's Wort) within 4 weeks prior to Visit 1 or planning to start during the study period.
  13. Disease such as coeliac disease, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, gastroesophageal reflux disease (GERD) that by the investigator's judgement, could interfere with the intestinal barrier function or have undergone significant gastrointestinal surgery (appendectomy and cholecystectomy acceptable).
  14. Participants consuming prebiotics (containing fructans, galacto-oligosaccharides, psyllium husk, inulin as main component), or probiotics within last 4 weeks prior to Visit 1.
  15. Participants consuming GABA or glutamate supplements, or any other supplements that are thought to directly affect digestive health and mental well-being within 4 weeks prior to Visit 1 which in the opinion of the investigator, impact the study outcomes.
  16. Participants with a current history of drug (including illicit drug) and /or alcohol abuse at the time of enrolment.
  17. Has received treatment involving experimental supplements in the past 4 weeks, at the discretion of the investigator.
  18. Major changes in lifestyle (i.e., diet, dieting, exercise level, travelling, supplements) for duration of the study.
  19. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
  20. Any Participant who is an employee of the study site or an Atlantia Clinical Trials employee or their immediate family member or a member of their household.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) Total Score from baseline to end of intervention | 4 weeks
  The PSS is a self-reported measure of stress. The questions in this scale ask about participants feelings and thoughts during the last month. Respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. It is a 10-item questionnaire and has a total score which correlates with one of three score categories (low stress [0-13], moderate stress [14-26]and high stress

SECONDARY OUTCOMES:
Profile of Mood States Questionnaire (POMS) | 4 weeks
  POMS is a psychological rating scale used to assess transient, distinct mood states. It has seven subscales, including tension-anxiety, depression-dejection, anger-hostility, vigour-activity, fatigue-inertia, confusion-bewilderment, and friendliness. The researcher combines these scores to provide an overall measure called total mood disturbance.
Plasma GABA levels | 4 weeks
  Levels of Gamma-aminobutyric Acid in plasma
Salivary cortisol awakening response | 4 weeks
  c) Salivary cortisol awakening response at T0, T30, T45, T60 minutes
VAS scale on acute effects on stress | 30 hours
  The VAS (visual analogue scale) is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the parameter measured, e.g., the left end = no stress, and the right end = extreme stress
Faecal GABA quantification | 4 weeks
  Absolute quantification

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Prof, Principal Investigator — Atlantia Clinical Trials
Locations (1):
- Atlantia Clinical Trials, Cork, Co Cork, Ireland

IPD SHARING:
Plan to Share IPD: No